CLINICAL TRIAL: NCT03009305
Title: Cerebral Oxygen Saturation, Mean Systemic Filling Pressure and Haemodynamic Effects of PEP and CPAP in Lower Body Negative Pressure
Brief Title: Cerebral Oximetry in Lower Body Negative Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Aslak Landsverk, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/3995
Record Dates: First submitted 2015-10-26; First posted 2017-01-04 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia | interventions — Lower Body Negative Pressure; Continuous Positive Airway Pressure; Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lower body negative pressure (Experimental): Single-arm, lower body negative pressure, continuous positive airway pressure, positive expiratory pressure.
  Interventions: Other: Lower body negative pressure; Device: Continuous positive airway pressure; Device: Positive expiratory pressure

INTERVENTIONS:
Other: Lower body negative pressure — Model of hypovolemia: Lower body negative pressure down to -80 mmHg (maximum).
Device: Continuous positive airway pressure — CPAP of 0, 5 and 10 cm water (H2O).
  Other Names: CPAP
Device: Positive expiratory pressure — PEP of 0, 5 and 10 cm H2O.
  Other Names: PEP

SUMMARY:
The study aims to describe hemodynamic effects of lower body negative pressure (LBNP).

1. If and how changes in cerebral oxygen saturation (StO2) measured by near infrared spectroscopy (NIRS) relate to changes in blood flow in the carotid arteries during progressive LBNP.
2. If and how mean systemic filling pressure (MSFP) can be measured by brief occlusion of blood flow to an arm and if this relates to LBNP-level.
3. If and how pulse pressure variations and photoplethysmographic amplitude variations during positive expiratory pressure (PEP) and continuous positive airway pressure (CPAP) relate to LBNP-level.

DETAILED DESCRIPTION:
20 healthy volunteers will be included. The study protocol consists of two parts.

1. LBNP is applied stepwise (20 mmHg increments). At each LBNP-level, after 2 min stabilization, blood flow in internal and external carotid arteries is measured. Thereafter, MSFP is measured. LBNP is applied to -80 mmHg, but terminated sooner if the subject experiences signs of decompensation.

   Changes in cerebral StO2 will be related to relative changes in blood flow in the carotid arteries. After these measurements, blood flow to one arm will be occluded for 30 s. Venous pressure measured in an antecubital vein approximates MSFP. This will be related to volume status (LBNP-level and stroke volume reduction).
2. LBNP is applied stepwise (20 mmHg increments). At each LBNP-level, after 2 min stabilization, PEP and CPAP are applied at 0, 5 and 10 cmH20. LBNP is applied to -80 mmHg, but terminated sooner if the subject experiences signs of decompensation.

Flow in carotid arteries is measured by ultrasound/Doppler. Skin blood flow in the forehead measured by laser Doppler flowmetry and transcutaneous oxygen saturation.

If possible, blood flow velocity in a. cerebri media will be measured by transcranial Doppler.

Central venous pressure will be approximated by measuring pressure in the left subclavian vein ("half-way" catheter).

Cardiac stroke volume will be measured by suprasternal Doppler. Expiratory carbon dioxide (CO2) will be measured and recorded. Acral skin photoplethysmography performed using proprietary and custom-made photoplethysmographs.

Arterial blood pressure approximated by finger volume-clamp method.

The measurements above will be used for analyses of possible physiological mechanisms and post-hoc analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (informed consent)

Exclusion Criteria:

* Disease/physical condition limiting normal physical activity or requiring medication (except allergies/contraceptives)
* History of syncope (except with obvious vasovagal etiology)
* Cardiac arrhythmia
* Pregnancy
* Skin infections in the elbow crease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
StO2 (tissue oxygen saturation). | Approximatrly 30 min: From start LBNP (lower body negative pressure) exposure to 5 min after end LBNP.
  Association between cerebral StO2 and flow in a. carotis interna.

SECONDARY OUTCOMES:
MSFP, mean systemic filling pressure (arm venous pressure during vascular occlusion). | Approximatrly 30 min: From start LBNP (lower body negative pressure) exposure to 5 min after end LBNP.
  Association between MSFP and volume status.
Dynamic variables and PEP (positive expiratory pressure)/CPAP (continuous positive airway pressure) | Approximatrly 30 min: From start LBNP (lower body negative pressure) exposure to 5 min after end LBNP.
  Association between dynamic variables during PEP/CPAP and volume status. Dynamic variables (variations in arterial pressure and photoplethysmographic waveforms with respiration) are calculated during with PEP and CPAP during hypovolemia (lower body negative pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Svein Aslak Landsverk, M.D., PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway